CLINICAL TRIAL: NCT05772520
Title: A Randomized, Double-blinded, Placebo-controlled, Multicenter Phase 2 Study Evaluating the Efficacy and Safety of TLL018 in Participants With Moderate-to-severe Plaque Psoriasis
Brief Title: The Efficacy and Safety of TLL018 in Moderate-to-severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Highlightll Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TLL018-205
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2023-09

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 2 (Experimental): TLL018 tables, 20 mg 1piece,BID
  Interventions: Drug: TLL018 tablets
- Cohort 3 (Experimental): TLL018 tables, 40 mg 1piece,BID
  Interventions: Drug: TLL018 tablets
- Cohort 4 (Experimental): placebo, 1piece,BID
  Interventions: Drug: TLL018 tablets

INTERVENTIONS:
Drug: TLL018 tablets — oral tablets administered 20 mg BID and 40 mg BID for 12 weeks
  Other Names: TLL018 Placeboes

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blinded, parallel dose group, placebo-controlled, dose-ranging study to evaluate the efficacy and safety of 2 doses of TLL018 as therapy in approximately 90 participants with moderate-to-severe PP.

ELIGIBILITY:
Inclusion Criteria:

1. Are between the ages of 18 and 75 years, inclusive, at time of informed consent.
2. Capable of giving informed consent and complying with study procedures.
3. Willing and able to adhere to study restrictions.
4. Laboratory and medical history parameters within the protocol defined ranges.
5. Normal renal function (>90 mL/min/1.72 m2) or mild renal impairment (Stage 2 mild chronic kidney disease glomerular filtration rate [GFR] = 60 to 89 mL/min/1.73 m2) as determined by central laboratory.
6. Body mass index (BMI) of 18.0 to 35.0 kg/m2 inclusive.
7. Have had a diagnosis of moderate-to-severe PP for at least 6 months prior to Baseline.
8. Participants with moderate-to-severe PP covering ≥10% body surface area (BSA), with a Psoriasis Area and Severity Index (PASI) ≥12 and a static Physician's Global Assessment (PGA) score ≥3 at Baseline.
9. Participants with plaque psoriasis who are systemic treatment naïve or have received at least one of the conventional anti-psoriasis treatments such as acitretin, phototherapy, methotrexate, cyclosporine, apremilast, or biologic therapy (anti-TNF or anti-IL-12/17/23).
10. Participants who are candidates for systemic treatment for psoriasis at the discretion of the Investigator.
11. Must agree to avoid prolonged exposure (> 15 minutes) to the sun and avoid use of tanning booths or other ultraviolet light sources during the study.
12. Female participants of childbearing potential (See Section 10.4.1 definition of Woman of Childbearing Potential - WOCBP) must have a negative serum human chorionic gonadotropin (hCG) at Screening, and meet one of the following criteria:

    1. Using a medically acceptable form of birth control (Appendix 4) for at least 1 month prior to Screening and 3 months after the last dose of study drug (e.g., hormonal contraceptives [oral, patch, injectable or vaginal ring], implantable device [implantable rod or intrauterine device], bilateral tubal occlusion/tubal ligation, azoospermic partner).
    2. Abstinence as a form of birth control is generally not permitted during the study with the exception of participants who practice abstinence as a preferred and usual lifestyle style choice. The Investigator must confirm that abstinence is still in accordance with the participant's lifestyle at regular intervals throughout the study.
13. Male participants with female partners of childbearing potential must agree to use condoms for the duration of the study and until 13 weeks after administration of the study intervention and must refrain from donating sperm for this same period. In addition, his female partner should agree to use a highly effective method of birth control per Appendix 4 or an additional barrier form of birth control (e.g., diaphragm, cervical cap, spermicide, or sponge).)
14. Ability to swallow and retain oral study intervention.
15. Participants must have completed their coronavirus disease 2019 (COVID-19) vaccination in accordance with the latest CDC guidelines, which is based on previous vaccination history. Please reference COVID-19 vaccination guidance for individuals who are moderately or severely immunocompromised (Clinical Guidance for COVID-19 Vaccination | CDC).

    1. Previous Pfizer-BioNTech, Moderna or Novavax: Must have previously received at least a 1st and 2nd dose, then must have received an updated formulation according to the CDCs dosing requirements; or
    2. Novavax or Johnson and Johnson's Janssen: Must have previously received 1 or more doses in combination with any original monovalent or bivalent COVID-19 vaccine doses, then must receive an updated formulation according to the CDCs vaccination guidelines.

       ...

Exclusion Criteria:

1. Pregnant or nursing women.
2. Past history of gastrointestinal perforation, history of peptic ulcers and/or regular use of NSAIDs.
3. History of chronic alcohol or drug abuse within 6 months prior to Screening as determined by the Investigator based on medical history and patient interview.
4. Current or recent history of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, metabolic, endocrine, pulmonary, cardiovascular, neurologic, or psychiatric disease.
5. Current and/or recent history (<30 days prior to Screening and/or <45 days prior to randomization) of a clinically significant viral, bacterial, fungal, parasitic, or mycobacterial infection.
6. Subject is currently being treated with or has received strong cytochrome P450 3A (CYP3A4) inhibitors, such as itraconazole, within 4 weeks prior to Baseline (Day 0).
7. Any history of malignancies, except for non-recurrent basal cell skin cancer, squamous cell skin cancer, and cervical cancer in situ that are considered to be cured.
8. Tests positive for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV). For Hepatitis B all subjects will undergo testing for Hepatitis B Surface Antigen (HBsAg) and Hepatitis B Core Antibody (HBcAb). Subjects who are HBsAg positive are not eligible for the study. Subjects who are HBsAg negative and HBcAb positive will subsequently need testing for Hepatitis B virus deoxyribonucleic acid (HBV DNA) and if HBV DNA negative may be enrolled in the study; if HBV DNA is positive, the subject is not eligible for the study. Positive hepatitis C virus result is defined as having a positive hepatitis C antibody test with a positive confirmatory hepatitis C polymerase chain reaction test.
9. Recent exposure to active tuberculosis (TB). Current evidence of active TB or current evidence of latent TB. Participants with positive TB test (e.g., QuantiFERON) that have been treated for latent TB. A borderline QuantiFERON test should be repeated. If still indeterminant, then a chest x-ray may be performed (positive chest x-ray is exclusionary).
10. History of unexplained syncope, symptomatic hypotension, or hypoglycemia.
11. Abnormal D-dimer levels in conjunction with clinical or current and past thrombotic disease.
12. Participants with uncontrolled hypertension, uncontrolled diabetes, untreated or uncontrolled hyperlipidemia (fasting blood triglycerides >500 mg/dL and fasting cholesterol >250 mg/dL).
13. History of any significant cardiac event (e.g., myocardial infarction) within 6 months prior to Screening, including:

    1. History of long QTc syndrome; history or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant.
    2. History of unstable ischemic heart disease or uncontrolled hypertension.
    3. Current Class 3 or 4 heart failure per the New York Heart Association Functional Classification.
    4. Screening and/or Baseline QTcF > 450 msec for males and > 470 msec for females, confirmed by triplicate ECG.
14. Participants with history of thrombosis and/ or thromboembolism, or associated risk factors (e.g., inherited thrombophilias, etc.).
15. Donated or lost >500 mL of blood in the previous 3 months.
16. Participants with chronic kidney disease with eGFR <60 mL/min/1.73 m2.
17. Participants with moderate-to-severe hepatic impairment (i.e., Child-Pugh Class B and C).
18. Major surgery within 3 months prior to Screening or participant has a planned major surgery during the course of the study.
19. Participants with any of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study-specific laboratory and confirmed by a single repeat, if deemed necessary:

    * Hemoglobin <100 g/L
    * White blood cell (WBC) count of <3.0 × 109/L
    * Platelet count of <80 × 109/L
    * Absolute neutrophil count of <1.5 × 109/L
    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values greater than 3 times the ULN
20. Any uncontrolled clinically significant laboratory abnormality that would affect interpretation of study data or the participant's participation in the study.
21. Previous or current autoimmune diseases (e.g., RA, systemic lupus erythematosus, IBD, scleroderma, inflammatory myopathy, mixed connective tissue disease overlap syndrome, etc.). Note, psoriatic arthritis patients are allowed.
22. Other types of psoriasis (such as erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, drug-induced psoriasis).
23. Current enrollment in another study intervention protocol or experimental treatment within 30 days or five half-lives (whichever is longer).
24. Received any topical therapy that can affect psoriasis (including topical use of moderate-strong glucocorticoids, retinoids, vitamin D3 derivatives, salicylic acid, anthracene, etc.) within 2 weeks of first study intervention. Low potency topical steroids are permitted for sensitive areas only (e.g., face, axillae, genitalia). Bland emollients without urea or α or β-hydroxy acids are permitted.
25. Use of phototherapy (including photochemotherapy, ultraviolet therapy, tanning bed self-therapy, etc.) within 4 weeks of first study intervention.
26. Use of systemic oral therapy that can affect psoriasis (including but not limited to glucocorticoids, retinoids, cyclosporine, methotrexate and apremilast) within 4 weeks of first study intervention.
27. Received intravenous corticosteroids within 4 weeks of first study intervention.
28. Use of antimalarial drugs, interferon-α, lithium and beta-blockers within 4 weeks of first study intervention.
29. Use of Chinese or herbal medicine treatment of psoriasis within 2 weeks of first study intervention.
30. Prior to randomization, washout periods of the following biologics are required: etanercept ≥28 days; any s.c. mAb targeting TNF (eg., infliximab, adalimumab, certolizumab) >3 months; ustekinumab or drugs that specifically target IL-23>6 months; secukinumab, ixekizumab, bimekizumab, brodalumab or other IL-17 antagonists >6 months; any other anti-psoriasis treatments not listed within 5 half-lives. Topical JAK inhibitors should have a washout period > 2 weeks.
31. Prior use of three or more biologic therapies.
32. Use of natalizumab and other drugs that regulate B or T cells within 12 months of first study intervention, such as rituximab, alemtuzumab, and abatacept.
33. Participants who have received live vaccines within 2 months prior to first study intervention or plan to receive live vaccines during the study period. Non-live-attenuated vaccines (e.g., ribonucleic acid [RNA]-based vaccines, inactivated adenovirus-based vaccines, protein-based vaccines), including non-live-attenuated vaccines or boosters for coronavirus disease 2019 (COVID-19) during the study are allowed.
34. Participants who have received COVID-19 vaccines within 2 weeks of Baseline or participants who plan to receive COVID-19 vaccines during the study period (boosters are allowed).
35. Previously not completed COVID-19 vaccination in accordance with the CDC guidelines.
36. Participants who are allergic to any component of the study intervention or who are at risk for allergy as determined by the Investigator during the study.
37. Any condition for which the Investigator considers the participant inappropriate to participate in this study.

    ....

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
proportion of participants achieving PASI-75 | Week12
  A patient was a responser if a minimum 75% PASI improvement from Baseline was achieved including measure of the average redness (erythema), thickness (induration), and scaliness (scaling)
  In calculating the PASI, severity is determined by dividing the body into four regions: head (h), upper extremities (u), trunk (t), and lower extremities (l).Each of these areas is assessed separately for erythema, induration, and scaling, which are rated on a scale of 0 (none) to 4 (very severe). Extent of psoriatic involvement is graded as follows:
  0 = no involvement
  1. = 1% to 9%
  2. = 10% to 29%
  3. = 30% to 49%
  4. = 50% to 69%
  5. = 70% to 89%
  6. = 90% to 100%. PASI = 0.1 (Eh + lh + Sh) Ah + 0.2 (Eu + lu + Su) Au + 0.3 (Et +lt + St) At + 0.4 (El +ll +Sl) Al

SECONDARY OUTCOMES:
Proportion of participants achieving PGA score of 0 or 1 | From week 4 to Weeks 12
  A patient was a responser if PGA score of 0 or 1 condition was reached, as listed: (0 Clear) No signs of psoriasis, but post-inflammatory discoloration may be present; (1 Almost clear): Only minimal plaque elevation, scaling, and erythema.
Proportion of participants achieving PASI-75 (except Week 12) | From week 4 to Weeks 12(except Week 12)
  A patient was a responser if a minimum 75% PASI improvement from Baseline was achieved including measure of the average redness (erythema), thickness (induration), and scaliness (scaling)
  In calculating the PASI, severity is determined by dividing the body into four regions: head (h), upper extremities (u), trunk (t), and lower extremities (l).Each of these areas is assessed separately for erythema, induration, and scaling, which are rated on a scale of 0 (none) to 4 (very severe). Extent of psoriatic involvement is graded as follows:
  0 = no involvement
  1. = 1% to 9%
  2. = 10% to 29%
  3. = 30% to 49%
  4. = 50% to 69%
  5. = 70% to 89%
  6. = 90% to 100%. PASI = 0.1 (Eh + lh + Sh) Ah + 0.2 (Eu + lu + Su) Au + 0.3 (Et +lt + St) At + 0.4 (El +ll +Sl) Al
Proportion of participants achieving PASI-90 | From week 4 to Weeks 12
  A patient was a responser if a minimum 90% PASI improvement from Baseline was achieved including measure of the average redness (erythema), thickness (induration), and scaliness (scaling)
  In calculating the PASI, severity is determined by dividing the body into four regions: head (h), upper extremities (u), trunk (t), and lower extremities (l).Each of these areas is assessed separately for erythema, induration, and scaling, which are rated on a scale of 0 (none) to 4 (very severe). Extent of psoriatic involvement is graded as follows:
  0 = no involvement
  1. = 1% to 9%
  2. = 10% to 29%
  3. = 30% to 49%
  4. = 50% to 69%
  5. = 70% to 89%
  6. = 90% to 100%. PASI = 0.1 (Eh + lh + Sh) Ah + 0.2 (Eu + lu + Su) Au + 0.3 (Et +lt + St) At + 0.4 (El +ll +Sl) Al

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Cahaba, Birmingham, Alabama
  - Moy, Fincher, Chipps, Beverly Hills, California
  - Metropolis Derm, Los Angeles, California
  - Amicis Research Center, Northridge, California
  - Integrative Skin, Sacramento, California
  - Skin Surgical, San Diego, California
  - Life Clinical Trials, Coral Springs, Florida
  - Palm Beach, DeLand, Florida
  - D&H Doral Research Center LLC, Doral, Florida
  - Sweet Hope Research Specialty, Inc, Hialeah, Florida
  - CNS - Jacksonville, Jacksonville, Florida
  - CNS - Orlando SODO, Jacksonville, Florida
  - Altus Research, Lake Worth, Florida
  - Anchor Medical Research, LLC (Core Clinical Trials), Miami, Florida
  - Reserka Research, Miami, Florida
  - ForCare Medical (CenExcel), Tampa, Florida
  - Integrated Clinical Trial Services, Inc, Des Moines, Iowa
  - IMA Clinical Research, Monroe, Louisiana
  - Lawrence Green, Rockville, Maryland
  - Metro Boston, Brighton, Massachusetts
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - Revival Research Institute, Troy, Michigan
  - Grekin Skin, Warren, Michigan
  - Minnesota Clinical Study Center, New Ulm, Minnesota
  - Mount Sinai, New York, New York
  - Sadick Research Group, New York, New York
  - Remington-Davis, Inc., Columbus, Ohio
  - DermDox, Sugarloaf, Pennsylvania
  - CRCC, Charleston, South Carolina
  - Dermatology Associates of Knoxville, Knoxville, Tennessee
  - Derm Research, Austin, Texas
  - Studies in Dermatology, LLC, Cypress, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Progressive Clinical Research Group, Inc., San Antonio, Texas
  - Acclaim, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No